CLINICAL TRIAL: NCT00404755
Title: Dichotic Listening as a Predictor of Medication Response in Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #5294R; IRB 5294R (Other Grant/Funding Number: There is no grantor or funder)
Record Dates: First submitted 2006-11-28; First posted 2006-11-29 (Estimated); Results first posted 2018-03-15 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-03

CONDITIONS: Major Depressive Disorder; Dysthymia
Keywords: Depression
MeSH Terms: conditions — Depressive Disorder, Major; Dysthymic Disorder; Depression | interventions — Escitalopram; Bupropion; Imipramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- escitalopram (Experimental): escitalopram 10 mg/d for 1 week, then increasing by 10 mg/week if tolerated and not remitted to maximal dose of 40 mg/d
  Interventions: Drug: escitalopram
- bupropion (Experimental): bupropion extended release (XL) 150 mg/d for a week, then 300 mg/d for a week and then 450 mg/d; all dose increases if tolerated and not remitted
  Interventions: Drug: bupropion
- imipramine (Experimental): imipramine 50 mg/d increasing twice weekly by 50 mg/increase to 200 mg/d, then by 50 mg/week to a maximum dose of 300 mg/d; all dose increases if tolerated and not remitted
  Interventions: Drug: imipramine

INTERVENTIONS:
Drug: escitalopram — Escitalopram: wk 1: 10 mg/d; wks 2-3: 20 mg/d; wk4: 30 mg/d; wks 5-6: 40 mg/d
  Other Names: Lexapro.
  Arms: escitalopram
Drug: bupropion — bupropion XL 150 mg/d increasing as tolerated and not remitted by 150 mg/d to maximal dose of 450 mg/d
  Other Names: Wellbutrin
  Arms: bupropion
Drug: imipramine — imipramine 50 mg/d increasing twice weekly by 50 mg/increase to 200 mg/d, then 50 mg increase/week to 300 mg/d; all dose increases if tolerated and not remitted
  Other Names: Tofranil
  Arms: imipramine

SUMMARY:
This study will recruit 100 depressed patients to test whether the previous finding of an association between treatment response (with treatment groups including placebo, imipramine, and fluoxetine) and preferences of hemispheric laterality in perceptual processing are also found with a different type of commonly used anti-depressant, bupropion.

DETAILED DESCRIPTION:
Preliminary data suggest that depressed patients with increased left hemispheric laterality of perceptual processing are unlikely to improve during 6 weeks' treatment with placebo, while being very responsive to either imipramine or fluoxetine. Depressed patients who do not show evidence of poor right hemispheric functioning respond significantly more often to placebo than those with poor right hemispheric functioning , and do not show an advantage of drug over placebo. 100 patients will be tested with verbal and nonverbal dichotic tests, and then treated sequentially with bupropion, escitalopram, and imipramine. Preferential hemisphere for auditory processing will be correlated with treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Ages between 18-65
2. Meets Diagnostic and Statistical Manual, Fourth Edition (DSM-IV) criteria for current Major Depression, Dysthymia or Depression Not Otherwise Specified

Exclusion Criteria:

1. Known Hearing impairment
2. Active suicidal ideation (history of suicide attempts will be evaluated on a case by case basis).
3. Hamilton Rating Scale for Depression (HAMD), 21-item total score >20
4. Current (past 6 months)alcohol and/or drug abuse or dependence
5. Medical condition likely to require intervention contraindicated with study medication (e.g., known arrhythmia likely to be exacerbated by Imipramine)
6. Bipolar I
7. Psychosis
8. Non-response to adequate trial of study medication (i.e., > or = 4 weeks on > or = bupropion 300mg/d, escitalopram 30mg/d, or imipramine 200mg/d)
9. Premenopausal women not using known effective birth control
10. Not currently depressed (whether considered due to current treatment or not)
11. History of seizure, seizure disorder, anorexia nervosa, or bulimia
12. Left-handed -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan W. Stewart, M.D., Principal Investigator — New York State Psychiatric Institute; Gerard Bruder, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Depression Evaluation Service official website — http://www.depression-nyc.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 7/24/2006 - 4/7/2008 Recruitment Location: outpatient research clinic
Pre-assignment Details: Patients had to have not taken psychotropic medication for at least two weeks (no fluoxetine for at least 5 weeks) and had to produce a urine negative for commonly abused substances. Current use of psychotropic medication or a positive urine toxicology screen would abort further study participation.
Groups:
- Bupropion: this was the initial treatment given to all patients except one who was ineligible for bupropion and received escitalopram
  bupropion extended release (XL) 150 mg/d for a week, then 300 mg/d for a week and then 450 mg/d; all dose increases if tolerated and not remitted
  bupropion: bupropion XL 150 mg/d increasing as tolerated and not remitted by 150 mg/d to maximal dose of 450 mg/d
Period: Phase I (Bupropion)
Arm/Group | Bupropion
Started | 17 (3 went directly into Phase II (intolerant of bupropion), 1 withdrew consent and 4 did not return)
Completed | 13
Not Completed | 4
Not completed — Adverse Event | 3
Not completed — Other | 1
Period: Phase II (Escitalopram)
Arm/Group | Bupropion
Started (Escitalopram 10mg/d RX to those not improved in PhaseI for 1 wk, then to 20, maximal dose of 40mg/d) | 11
Completed | 9
Not Completed | 2
Not completed — Lost to Follow-up | 2
Period: Phase III (Imipramine)
Arm/Group | Bupropion
Started (imipramine 50mg/d increasing twice wkly by 50mg upto 200mg/d, to maxdose of 300mg/d II nonremitters) | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Bupropion: bupropion XL 150 mg/d for a week, then 300 mg/d for a week and then 450 mg/d; all dose increases if tolerated and not remitted
  bupropion: bupropion XL 150 mg/d increasing as tolerated and not remitted by 150 mg/d to maximal dose of 450 mg/d
Arm/Group | Bupropion
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Scale (HAM-D)
Description: Hamilton Depression Scale, 21 item version Summary of all 21 items and higher score means worse depression. Scores range from 0 to a maximum of 63.
Time Frame: 6 weeks or last visit in Phase
Population: Participants were included if they were given that medication
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupropion | Escitalopram | Imipramine
Number analyzed (Participants) | 17 | 10 | 3
units on a scale | 11.2 (7.9) | 9.7 (6.4) | 11.3 (8.1)

2. Secondary Outcome: Clinical Global Impression Scale (CGI)
Description: The CGI is a standard measure of global psychopathology. CGI-severity scores rated on a 7-point scale, with the severity of illness scale using a range of responses from
  1 (normal) through to 7 (amongst the most severely ill patients). CGI-improvement scores range from 1 (very much improved) through to 7 (very much worse).
Time Frame: 6 weeks or last visit in Phase
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupropion | Escitalopram | Imipramine
Number analyzed (Participants) | 17 | 11 | 3
units on a scale | 2.65 (1.12) | 2.73 (1.10) | 2.67 (0.58)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: 6 weeks
Arm/Group | Escitalopram | Bupropion | Imipramine
Serious Adverse Events (participants affected / at risk) | 0/11 | 1/17 | 0/3
Other Adverse Events (participants affected / at risk) | 10/11 | 10/17 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram (N=11) | Bupropion (N=17) | Imipramine (N=3)
allergic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) — rash resolved within 48 hours of discontinuing medication
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram (N=11) | Bupropion (N=17) | Imipramine (N=3)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) — queasy stomach
anorgasmia (Reproductive system and breast disorders) | 5 (5) | 0 (0) | 0 (0) — delayed, inability to reach orgasm
headache (General disorders) | 1 (1) | 3 (3) | 0 (0) — headache
overstimulatioin (General disorders) | 0 (0) | 2 (2) | 0 (0) — too "revved up"
insomnia (General disorders) | 1 (1) | 3 (3) | 0 (0) — trouble sleeping
allergic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) — drug allergy
dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) — dry mouth
constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) — hard stool
a.m. grogginess (General disorders) | 0 (0) | 0 (0) | 1 (1) — feeling "drugged" in the morning
orthostatic hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) — dizziness on standing

LIMITATIONS AND CAVEATS:
This is an open (i.e., unblinded) study having small sample size

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No